CLINICAL TRIAL: NCT06975163
Title: Effectiveness of Mindfulness-Based Intervention in Reducing Stigma Stress Among Parents of Autistic Children: A Randomized Controlled Trial
Brief Title: Effectiveness of Mindfulness-Based Intervention in Reducing Stigma Stress Among Parents of Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN Ka Shing Kevin, Professor, Head of Department of Psychology, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-2021-0126
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Mindfulness; Stigma stress; Parents
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Stigma Stress Reduction (MBSSR) group (Experimental): Participants in the MBSSR group received a 4-week MBSSR program immediately after randomization. Participants completed the post-intervention assessment right after the intervention and the follow-up assessment one month after the intervention.
  Interventions: Behavioral: Mindfulness-Based Stigma Stress Reduction (MBSSR) program
- Waitlist control group (No Intervention): Participants in the waitlist control group waited for 4 weeks without the Mindfulness-Based Stigma Stress Reduction (MBSSR) program. Participants completed the post-intervention assessment and the follow-up assessment simultaneously with the MBSSR group. After completing the follow-up assessment, the waitlist control participants started the MBSSR program (equivalent to that of the MBSSR group).

INTERVENTIONS:
Behavioral: Mindfulness-Based Stigma Stress Reduction (MBSSR) program — The MBSSR program was developed by modifying elements from the Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT) programs to create a distinct mindfulness intervention targeted at alleviating stigma stress among parents of autistic children. This program consisted of four group sessions, each incorporating mindfulness practices, group discussions, and activities that helped participants apply mindfulness principles to their daily lives.
  Arms: Mindfulness-Based Stigma Stress Reduction (MBSSR) group

SUMMARY:
Autism Spectrum Disorder (ASD) is a lifelong neurodevelopmental condition that usually becomes apparent in early childhood. Those diagnosed with ASD commonly struggle with social communication and behavioral regulation, often facing widespread societal stigma across different cultures. This prejudice extends beyond the affected children to their parents, who are routinely subjected to baseless blame and viewed as incapable of proper parenting. Such persistent negative perceptions can foster profound emotional suffering and chronic stress linked to societal judgment.

To date, there are no empirically supported interventions specifically aimed at alleviating stigma-induced stress in parents of autistic children. Nevertheless, studies in related fields indicate that mindfulness-based strategies could offer a potential coping mechanism. Addressing this gap, the current research presents a newly developed 4-week Mindfulness-Based Stigma Stress Reduction (MBSSR) program tailored for these parents. Using a randomized controlled trial, participants were divided into an MBSSR group or a waitlist control group, with both undergoing standardized evaluations at three distinct time points.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a well-known neurodevelopmental condition that emerges in early childhood and continues into adulthood. Children with ASD frequently face social and behavioral difficulties, and research indicates that stigma surrounding autism is prevalent in many societies. These children are sometimes mistakenly perceived as deliberately unruly, resulting in social prejudice and exclusion. This stigma also affects their parents, who endure societal judgment due to their emotional and biological ties to their children. Parents may be wrongly blamed for passing on "faulty" genes or accused of causing their child's condition. Additionally, they are often labeled as incompetent caregivers and criticized for failing to properly handle their child's behavior. Prolonged exposure to such bias can trigger deep-seated shame and psychological distress, leading to persistent stress linked to stigma.

Although stigma-related stress significantly impacts parents of autistic children, there are currently no scientifically validated interventions specifically designed to help them manage it. However, studies in similar areas propose that mindfulness practices may help individuals deal with stigma-induced stress. To bridge this research gap, this study introduces a novel 4-week Mindfulness-Based Stigma Stress Reduction (MBSSR) program tailored for parents of children with autism in Hong Kong. Using a randomized controlled trial approach, participants were divided into either the MBSSR treatment group or a waitlist control group, with both groups undergoing standardized evaluations at three separate intervals.

ELIGIBILITY:
Inclusion Criteria:

* Having a child formally diagnosed with Autism Spectrum Disorder (ASD) under Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria by a registered medical practitioner
* Acting as the principal caregiver for the child
* Having the ability to read and write in Chinese
* Demonstrating the experience of stigma stress on the Family Stigma Stress Scale, defined as agreeing with item(s) that gauge perceived stigma harm and disagreeing with item(s) that evaluate perceived coping resources

Exclusion Criteria:

* Having participated in any mindfulness-based programs before
* Currently using psychiatric medications or receiving mental health services from professionals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Assessment in Stigma Stress on the Stigma Stress Scale at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The Stigma Stress Scale was utilized to assess perceived stigma harm and perceived coping resources on a 5-point scale where 1 indicated "strong disagreement" and 5 indicated "strong agreement".

SECONDARY OUTCOMES:
Change from Baseline Assessment in Well-being on the World Health Organization Well-Being Index at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The World Health Organization Well-Being Index was utilized to assess well-being on a 6-point scale where 0 indicated "at no time" and 5 indicated "all of the time".
Change from Baseline Assessment in Caregiving Gain on the Positive Aspects of Caregiving at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The Positive Aspects of Caregiving was utilized to assess caregiving gain on a 5-point scale where 1 indicated "disagree a lot" and 5 indicated "agree a lot".
Change from Baseline Assessment in Caregiving Burden on the Zarit Burden Interview at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The Short Version of the Zarit Burden Interview was utilized to assess caregiving burden on a 5-point scale where 1 indicated "never" and 5 indicated "nearly always".
Change from Baseline Assessment in Mindful Parenting on the Interpersonal Mindfulness in Parenting Scale at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The Interpersonal Mindfulness in Parenting Scale was utilized to assess mindful parenting on a 5-point scale where 1 indicated "never true" and 5 indicated "always true".
Change from Baseline Assessment in Child Autistic Symptoms on the Childhood Autism Rating Scale at Post-Intervention Assessment and Follow-up Assessment | Before intervention, immediately after intervention, and one month after intervention
  The Childhood Autism Rating Scale was utilized to assess child autistic symptoms on a 4-point scale where 1 indicated "normal" and 4 indicated "severely abnormal".

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ka Shing Chan, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No